CLINICAL TRIAL: NCT01379183
Title: Magnetic Resonance (MR) Evaluation of the Effect of Erythromycin Upon Gastric and Small Bowel Motility
Brief Title: Using Magnetic Resonance (MR) to Understand the Effect of Erythromycin on Bowel Motility
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeff Fidler, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10-004869; P01DK068055 (NIH)
Record Dates: First submitted 2011-06-15; First posted 2011-06-23 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Healthy; Men; Women; No known gastrointestinal disease; Aged between 18-70 years
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Erythromycin; Water; Sodium Chloride; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Active Comparator): Erythromycin 200 mg i.v. suspension, Barium Sulfate Solution, and Magnetic Resonance Imaging
  Interventions: Drug: Erythromycin; Procedure: Magnetic Resonance Imaging; Other: Barium Sulfate Solution
- Placebo (Placebo Comparator): Matching placebo i.v. suspension, Barium Sulfate Solution, and Magnetic Resonance Imaging
  Interventions: Drug: Placebo; Procedure: Magnetic Resonance Imaging; Other: Barium Sulfate Solution

INTERVENTIONS:
Drug: Erythromycin — 200 mg suspension
  Other Names: Erythromycin suspension
  Arms: Erythromycin
Drug: Placebo — 200 mg suspension
  Other Names: Water in 0.9% Sodium Chloride
  Arms: Placebo
Procedure: Magnetic Resonance Imaging — An MR enterography procedure uses magnetic resonance imaging (MRI) technology to obtain detailed images of the small bowel.
  Other Names: MRI; Magnetic Resonance Enterography
Other: Barium Sulfate Solution — Participants will be given a low concentration of barium sulfate solution (1350 mL) prior to the MRI procedure. Barium sulfate is a radiopaque agent. Radiopaque agents are used to help diagnose certain medical problems. Since radiopaque agents are opaque to (block) x-rays, the areas of the body in which they are localized will appear white on the x-ray film. This creates the needed distinction, or contrast, between one organ and other tissues. The contrast will help the doctor see any special conditions that may exist in that organ or part of the body.
  Other Names: VoLumen

SUMMARY:
Magnetic Resonance Imaging (MRI) has proven to be a valuable imaging technique for suspected small bowel disease. This technique depends, in part, on adequate distension of the small bowel. This is accomplished by administering large volumes of a non-absorbable oral contrast material prior to the examination, which typically produces excellent distension of the distal small bowel and stomach, but poor distension of the proximal small bowel. Erythromycin is a common antibiotic that is known to promote stomach emptying and is used to treat diabetics with gastroparesis (poor stomach emptying.) The hypothesis of this study was that erythromycin will increase gastric emptying and hence improve small and large intestinal distention during MRI.

DETAILED DESCRIPTION:
Gastric, small, and large intestinal volumes were assessed with MRI after ingestion of a low concentration of barium sulfate solution (1350 mL) and randomization to erythromycin 200 mg i.v.) or placebo in 40 healthy volunteers. Magnetic Resonance Images of the abdomen were acquired with a torso phased array coil and a 1.5 tesla magnet.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult volunteers without known gastrointestinal disease
* Aged 18-70 years
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

* Known allergy to erythromycin;
* Use of drugs that have known contraindication with erythromycin (concomitant therapy with astemizole, cisapride, pimozide, or terfenadine)
* Corrected QT interval on EKG >460 msec
* Certain medications (i.e., theophylline, digoxin, oral anti-coagulant, benzodiazepine, 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors) will either be excluded from the study or, if medically safe, will be asked to discontinue the medication for 4 half-lives before beginning the study.
* Use of medications that alter GI motility e.g., narcotics, medications with significant anticholinergic effects
* Pregnant or breast-feeding females
* Known claustrophobia
* Known family history of sudden death or congenital QT prolongation
* Presence of pacemaker, internal defibrillator, or other non-MR compatible device
* Patients with known metal present within their abdomen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Fidler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 07/09/2011 - 03/13/2013 Location: Mayo Clinic, Rochester, Minnesota
Pre-assignment Details: There was no wash out or run-in period following participant enrollment.
Groups:
- Erythromycin: Erythromycin 200 mg i.v. suspension
- Placebo: Matching placebo i.v. suspension
Period: Overall Study
Arm/Group | Erythromycin | Placebo
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythromycin | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12.6) | 35 (13) | 35 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Gastric Volume
Description: A Magnetic Resonance (MR) enterography procedure uses magnetic resonance imaging (MRI) technology to obtain detailed images of the small bowel. MR images of the abdomen were acquired with a torso phased array coil and a 1.5 tesla magnet MRI. Gastric volumes were assessed with an axial 3D axial gradient echo sequence, which imaged the entire stomach in 13 seconds.
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 262 (52) | 718 (59)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Jejunal Volume
Description: The jejunum is the section of the small intestine between the duodenum and the ileum. A Magnetic Resonance (MR) enterography procedure uses magnetic resonance imaging (MRI) technology to obtain detailed images of the small bowel. Small bowel volumes were evaluated with 5 mm thick coronal slices using a fat-suppressed true fast imaging with steady state precession sequence while the participant held his or her breath.
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 450 (74) | 359 (43)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.27, ANCOVA

3. Secondary Outcome: Ileal Volume
Description: The Ileal is the terminal portion of the small intestine extending from the jejunum to the cecum. A Magnetic Resonance (MR) enterography procedure uses magnetic resonance imaging (MRI) technology to obtain detailed images of the small bowel. Small bowel volumes were evaluated with 5 mm thick coronal slices using a fat-suppressed true fast imaging with steady state precession sequence while the participant held his or her breath.
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 248 (30) | 248 (27)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.96, ANCOVA

4. Secondary Outcome: Colonic Volume
Description: A Magnetic Resonance (MR) enterography procedure uses magnetic resonance imaging (MRI) technology to obtain detailed images of the small bowel. Small bowel volumes were evaluated with 5 mm thick coronal slices using a fat-suppressed true fast imaging with steady state precession sequence while the participant held his or her breath.
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 190 (53) | 180 (36)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.71, ANCOVA

5. Secondary Outcome: Small Intestine Volume
Description: as for outcome 4
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 698 (99) | 607 (56)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.37, ANCOVA

6. Secondary Outcome: Small Intestine and Colon Volume
Description: as for outcome 4
Time Frame: Approximately 60 minutes after beginning ingestion of fluid volume
Measure: Mean (Standard Error); unit: mL
Arm/Group | Erythromycin | Placebo
Number analyzed (Participants) | 19 | 21
mL | 910 (66) | 781 (65)
Statistical Analysis 1: Comparison: Erythromycin vs Placebo; Test type: Superiority or Other; p = 0.12, ANCOVA

ADVERSE EVENTS:
Arm/Group | Erythromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes